CLINICAL TRIAL: NCT05228873
Title: Comparison of Quality of Life 3 Months After Discharge of the Mild and Moderate COVID-19 Patients With or Without Herbal Medicine (Shen Cao Gan Jiang Tang) in the Acute Stage
Brief Title: Comparison of Quality of Life After Discharge of the Mild and Moderate COVID-19 Patients With or Without Herbal Medicine
Status: Completed | Type: Observational
Sponsor: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Responsible Party: Principal Investigator, NGUYEN VAN DAN, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Other Study IDs: 838-9/HĐĐĐ-ĐHYD
Record Dates: First submitted 2022-02-05; First posted 2022-02-08 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: COVID-19 Pandemic; Quality of Life
MeSH Terms: conditions — COVID-19 | interventions — Asian ginseng

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Investigational arm: Patients take Shen Cao Gan Jiang Tang (Gan Cao Gan Jiang Tang with Ginseng), one bag of decoction (90ml) two times a day for 10 days plus the Standard of Care (SOC) for the treatment of COVID-19 acute stage based on the Vietnam Ministry of Health guideline at this time
  Interventions: Drug: Shen Cao Gan Jiang Tang (Gan Cao Gan Jiang Tang with Ginseng)
- • Controlled arm: Patient who receive the Standard of Care (SOC) for the treatment of COVID-19 acute stage based on the Vietnam Ministry of Health guideline at this time

INTERVENTIONS:
Drug: Shen Cao Gan Jiang Tang (Gan Cao Gan Jiang Tang with Ginseng) — Patients take Shen Cao Gan Jiang Tang (Gan Cao Gan Jiang Tang with Ginseng), one bag of decoction (90ml) two times a day for 10 days. Ingredients per formula (tang): 12 grams of honey-fried Radix Glycyrrhizae, 6 grams of Rhizoma Zingiberis (stir-baked), 6 grams of Panax Ginseng. The decoction of concentrated extract is packed into aluminum foil vacuum bag, 90ml per bag, 1 formula (tang) is equivalent to 2 bags. Patients use the decoction directly from the bag.
  Other Names: Sâm Thảo Can khương thang (Cam thảo Can khương thang gia Nhân sâm) - Vietnamese name
  Groups: Investigational arm

SUMMARY:
The purpose of this study is to see how the acute stage COVID-19 treatments by use of herbal medicine (Shen Cao Gan Jiang Tang) affect quality of life and symptoms at 3 months after hospital discharge.

DETAILED DESCRIPTION:
According to the theory of Traditional medicine, the patient will suffer damage to Qi and Fluid in the acute phase and lead to damaged Yin and Qi in the post COVID-19 period.

The Shen Cao Gan Jiang Tang has the effect of enhance the Protective Qi, generating Fluid, is applied to treat the mild and moderate COVID-19 in the acute phase in some hospitals in Ho Chi Minh City, Viet Nam. The hypothesis is that with the use of the Shen Cao Gan Jiang Tang, the Qi and Yin will reduce the damage, so that the patient has a better quality of life and fewer post COVID-19 symptoms compared with the standard of care group

ELIGIBILITY:
Inclusion Criteria:

* Patients able to understand and fill out a questionnaire
* From full 18 to 64 years old;
* Patients with the mild and moderate COVID-19 who used Shen Cao Gan Jiang Tang in the acute phase for intervention group.
* Participants enrolled in protocol NCT05055427.
* Voluntarily consented to participate in the study

Exclusion Criteria:

* Patient who are not able to complete 100% of the questionnaire Criteria for stopping the study
* The patient cannot be contacted after 04 calls, each call is at least 06 hours apart on the survey days.
* The patient does not want to continue participating in the study.

Ages: 18 Years to 64 Years | Sex: All
Age Groups: Adult
Study Population: The mild and moderate COVID-19 patients who used the Shen Cao Gan Jiang Tang in the acute phase
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
Quality of Life (QoL) questionnaire | 3 months
  Data will be collected by using the 36-Item Short Form Survey (SF-36) QoL instruments at 3 months after hospital discharge.

SECONDARY OUTCOMES:
Post COVID-19 symptoms | 3 months
  Number of patients (%) have the post COVID-19 symptoms at 3 months after hospital discharge. The post COVID-19 symptoms have included cough, shortness of breath, fatigue, headache, attention disorder, hair loss, loss of smell, loss of taste, rapid breathing after activity, joint pain

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen Van Dan, Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (1):
- University of Medicine and Pharmacy at Ho Chi Minh City, Ho Chi Minh City, Vietnam